CLINICAL TRIAL: NCT01011374
Title: Impact of Lucentis on Psychological Morbidity in Patients With Macular Edema and Neovascularization Secondary to Retinal Vein Occlusion
Brief Title: Impact of Lucentis on Psychological Morbidity in Patients With Retinal Vein Occlusion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Retina Associates of Cleveland, Inc (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Lawrence J. Singerman, MD, Retina Associates of Cleveland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4638s
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Venous Retinal Branch Occlusion; Central Retinal Vein Occlusion; Retinal Vein Occlusion; Depression
Keywords: Retinal vein occlusion; Ranibizumab; Lucentis; Depression
MeSH Terms: conditions — Retinal Vein Occlusion; Depression | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ranibizumab (Lucentis) — 0.5 mg, administered intravitreally every 4 weeks
  Other Names: Lucentis

SUMMARY:
This is a prospective, single-center, non-randomized clinical study on the impact of intravitreally administered ranibizumab (Lucentis) treatment on vision-related functioning and emotional well-being in subjects with central or branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Evidence of central retinal vein occlusion, defined as documented retinal hemorrhage into all four quadrants with dilated veins, or branch retinal vein occlusion, as documented on clinical exam
* Age 18 years or over
* Central macular edema on clinical exam as well as imaging with a central thickness of ≥ 250 microns
* Visual acuity ranging from 20/8000 to 20/40
* Media clarity and patient cooperation sufficient to allow adequate testing utilizing OCT and FA
* No previous treatment that might compromise or confound assessment of the study outcomes
* Ability to speak and read English

Exclusion Criteria:

* Acute illness or cognitive or other impairment that, in the opinion of the investigator, would interfere with study requirements
* Concurrent ocular conditions likely to significantly compromise vision and contribute the macular compromise
* History of grid/focal laser in the study eye
* History of vitreal surgery
* Previous treatment with triamcinolone acetonide in either eye
* Previous use of bevacizumab, pegaptanib, or ranibizumab in either eye
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
* History of cerebrovascular accident within 1 year prior to Day 0
* Inability to comply with study or follow-up procedures
* Any cognitive defect as a result of mental disease, previous injury, or disease process that may interfere with interpretation of study results
* Visual acuity better than 20/40
* Pregnancy (positive pregnancy test) or lactation
* Inadequate contraception in premenopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures are changes in the VFQ-25, GHQ-12, and PHQ-9 survey scores from baseline through 24 weeks. | 24 weeks

SECONDARY OUTCOMES:
Secondary outcome measures are change in macular edema measured by OCT and estimated by central retinal thickening and correlations between change in visual acuity, depression, and retinal findings such as neovascularization, rubeosis, and perfusion. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Singerman, MD, Principal Investigator — Retina Associates of Cleveland
Locations (1):
- Retina Associates of Cleveland, Cleveland, Ohio, United States